CLINICAL TRIAL: NCT04550182
Title: Evaluation of the Impact of the Repositioning Schedule Adapted to the Risk of Pressure Ulcer of Patients in Intensive Care Unit
Acronym: PROMESREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP180674; 2019-A02287-50 (Other: ANSM)
Record Dates: First submitted 2020-01-06; First posted 2020-09-16 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Pressure Ulcer; Ischemic; Ischemic Ulcer
Keywords: Intensive care unit; ICU; adult critical care patients; repositioning schedule; patient handling; practical nursing; nursing care; pressure ulcers; decubitus ulcers; pressure injury
MeSH Terms: conditions — Pressure Ulcer; Ischemia | interventions — Patient Positioning

STUDY DESIGN:
Intervention Model Description: To assess efficacy of a positioning schedule whose frequency of positioning is adapted every day to pressure ulcer risk assessed by Braden scale on the occurrence of pressure ulcer in adult ICUs, in comparison with the routine patients' management (without positioning schedule adapted on PU risk) at the 28th day, or when leaving ICU, or at death if it occurs before.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individual positioning schedule (Experimental): Pressure ulcer prevention cares are provided according to the positioning schedule for every patient.
  Interventions: Procedure: Positioning schedule
- Standard care (No Intervention): Pressure ulcer prevention cares are provided according to usual practice of the ICU. Frequency and modality of positioning applied to the patients are collected.

INTERVENTIONS:
Procedure: Positioning schedule — The Braden scale will be collected every morning. Patients' care will be friction and repositioning applied at a frequency defined by the Braden scale:
  6 ≥ Braden ≤ 8: alternate positioning every 2 hours 9 ≥Braden ≤ 13: alternate positioning every 4 hours 14 ≥ Braden ≤ 17: No alternative of the positioning required, but a friction and an evaluation of the cutaneous state every 6 hours.
  18 ≥Braden ≤ 23: No alternative of the positioning required, but a friction and an evaluation of the cutaneous state every 12 hours.
  Positioning will alternate semi-lateral decubitus at 30, semi-Fowler 30° -30°, half-sitting position 45° with elevation of the lower limbs.
  A medical prescription as part of the daily reassessed care will ensure the absence of absolute contraindication to the mobilization or contraindication to certain positions.Friction will be performed during repositioning.
  Other Names: Positioning; prevention of pressure ulcers; repositioning program
  Arms: Individual positioning schedule

SUMMARY:
Pressure ulcers represent a major health issue because of their high incidence and their important consequences. There is an important risk of pressure ulcer acquisition for ICU patients with acute organ failure(s).

Specific risk factors identified in ICU are immobility, which accentuates the effects of friction and shears, as well as mechanical ventilation and the use of vasopressors.

A repositioning schedule is a guideline for pressure ulcer prevention, but repositioning frequency remains unknown.

Adaptation of the repositioning schedule to pressure ulcer risk assessment using Braden scale should decrease the emergence of pressure ulcer. This could limit their important consequences for ICU patients which add to their brittle clinical condition (infection, increased length of stay, mortality…).

DETAILED DESCRIPTION:
This is a multicenter randomized controlled cluster, parallel open study. In order to avoid a contamination bias between groups, this trial will be randomized at the center level. This randomization will lead to the formation of 2 groups: a group of control centers (usual care) and a group of interventional centers (repositioning schedule).

A visit to set up the study will be carried out before the beginning of the inclusions. During this visit, a training course will be delivered to the caregivers of all the research centers on the risk assessment of pressure ulcers using the Braden scale, the evaluation of the skin condition, the identification of the stages of pressure and their management as well as the collection of data necessary for this study. In addition, the interventional group centers will receive training on the application of the repositioning schedule.

The risk assessment for pressure ulcers using the Braden scale will be performed daily in both groups. All patients participating in research with a Braden scale ≤ 17 will benefit from a pressure ulcer prevention mattress.

Usual care:

Within the control group, repositioning schedule frequencies and positioning will be done according to the habits of the service. The daily collection form present in the room will collect information concerning the care related to the positioning of the patient (length of treatment, frequency of positioning, type of positioning, any adverse events occurring during this care), the evaluation of the patients 'cutaneous status, duration of pressure ulcer care and evaluation of the Braden scale. The possible contraindications to the positioning of the patients will be informed by the doctors on the medical prescription according to the current practice.

Repositioning schedule:

Within the interventional group the repositioning schedule will be applied according to the risk of pressure ulcer evaluated daily by the Braden scale. A medical prescription, as part of the care, will attest to the absence of absolute contraindication or relative to the procedure of mobilization.

Depending on the result of the Braden scale, the repositioning schedule is defined as follows:

6 ≥ Braden ≤ 8: alternate positioning every 2 hours; 9 ≥Braden ≤ 13: alternate positioning every 4 hours; 14 ≥ Braden ≤ 17: No alternative of the positioning required, but a friction and an evaluation of the cutaneous state every 6 hours.

18 ≥Braden ≤ 23: No alternative of the positioning required, but a friction and an evaluation of the cutaneous state every 12 hours

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old without legal protection;
* Invasive or non-invasive mechanical ventilation;
* Inclusion in the first 48 hours following mechanical ventilation and in a maximum of 6 hours after 48 hours
* No pressure ulcer at the time of inclusion (according to EPUAP);
* Hospitalized in intensive care for less than 72 hours;
* Consent signed by the patient or in the event of the patient's temporary inability to express his or her wishes, consent will be obtained from a relative and signed by the patient as soon as possible; or in the absence of a relative, an emergency inclusion may be made; in this case a consent to proceed must be signed by the patient as soon as possible.

Exclusion Criteria:

* Patient admitted to intensive care unit for the multiple trauma management with spinal cord injury;
* Patient concerned by a medical decision to withhold/withdraw life sustaining therapies at the time of potential inclusion.
* Patient recruited in any other interventional research studying mobilization or positioning of the patient and/or pressure ulcer prevention and/or being in exclusion period of any other research if concerned;
* Patient already included once in the study
* Person without any health insurance scheme or not benefiting from a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1232 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The proportion of pressure ulcer at day 28 | Up to 28 days
  To assess the efficacy of a positioning schedule whose frequency of positioning is adapted every day to pressure ulcer risk assessed by the Braden scale and to the clinical state of the patient in adult ICUs, compared to usual PU prevention management (without schedule daily adapted to PU risk) at the 28th day, or when leaving ICU, or at death if it occurs before.
  Efficacy of the procedure will be measured by the proportion of pressure ulcer at day 28 or at ICU discharge or death if it occurs before.

SECONDARY OUTCOMES:
Tolerance of a repositioning schedule in adult intensive care unit | Up to 28 days
  Tolerance of the procedure will be appreciated by the proportion of adverse events that occurred during repositioning.
  The adverse events are:
  * accidental removal of invasive devices (intubation probe, catheter, drain, gastric tube, urinary catheter);
  * the occurrence of hemodynamic or respiratory instability ( Heart rate <40 or > 130 / min, Systolic Blood Pressure <90 mmHg, oxygen saturation <90%) necessitating stopping repositioning.
Impact of repositioning schedule on the length of hospitalization in intensive care unit | Up to 28 days
  Length of intensive care unit stay
Evaluate the applicability of a repositioning schedule and clinical barriers to patients' repositioning schedule | Up to 28 days
  Analysis of the correlation between the realization of the repositioning schedule and the characteristics of the patients, the SOFA and SAPS2 scores, the administration of support therapies (mechanical ventilation, vasoactive drugs, renal replacement therapy purification, ECCO2R, ECMO) and the medical and paramedical contraindications provided by caregivers and physicians on the daily collection form.
Risk factors for pressure ulcer on critically ill patients | Up to 28 days
  Identify the factors leading to the development of a pressure ulcer by completing a daily collection form.
Impact of a repositioning schedule on the time spent caring for alternate position procedure prevention in adult intensive care units | Up to 28 days
  Care time dedicated to the prevention in adult ICU evaluated by the positioning times in the care of positioning reported on the daily collection form.
Impact of a repositioning schedule on the management of bedsores in adult intensive care units | Up to 28 days
  Management of pressure ulcers in adult ICU evaluated by the number of caregivers involved in the care of positioning reported on the daily collection form.
Impact of a repositioning schedule on invasive care therapy for pressure ulcers | Up to 28 days
  Proportion of pressure ulcers requiring one of the following: surgical intervention, negative pressure wound therapy (VAC), antibiotic treatment;
total cost of the procedure and cost per pressure ulcer avoided | Up to 28 days
  Impact of the repositioning schedule on hospital costs and the occurrence of pressure ulcers will be compared through cost-effectiveness analysis and budget impact analysis. We will perform an analysis for staff cost and an analysis for the hospital cost per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Daisy Mehay, Degree Nurse in intensive care, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Réanimation Médico-chirurgicale. Hôpital Tenon, AP-HP, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No